CLINICAL TRIAL: NCT05320068
Title: Phase III,randomized,double-blinded Clinical Trial to Evaluate the Effectiveness and Safety of Oral Vancomycin Vs Placebo in the Prevention of Recurrence of C.difficile Infection in Patients Under Treatment with Systemic Antibiotic Therapy
Brief Title: Oral Vancomycin Vs Placebo in the Prevention of Recurrence of Clostridioides Difficile's Infection
Acronym: PREVAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Julia Orígüen (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Julia Orígüen, Julia Origüen Sabater, MD, PhD, Principal Investigator., Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PREVAN-ICD
Record Dates: First submitted 2022-03-22; First posted 2022-04-11 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Clostridioides Difficile Infection
Keywords: Vancomycin oral capsules
MeSH Terms: conditions — Clostridium Infections | interventions — Vancomycin

STUDY DESIGN:
Intervention Model Description: Proportion 2:1 in favour to the intervention arm
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): A group of patients will be treated with a blinded capsule that contains 125mg of vancomycin every 6 hours for 10 days.
  Interventions: Drug: Oral Vancomycin
- Placebo group (Placebo Comparator): A group of patients will be treated with a blinded capsule that contains a placebo every 6 hours for 10 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral Vancomycin — A blinded capsule that contains 125mg of vancomycin every 6 hours during 10 days.
  Arms: Intervention group
Drug: Placebo — A blinded capsule that contains no vancomycin every 6 hours during 10 days.
  Arms: Placebo group

SUMMARY:
A phase III randomized clinical trial in proportion 2:1 in favor of oral vancomycin (experimental treatment), multicentric, national, double-blinded, controlled with placebo. The main objective is to evaluate the effectiveness of treatment with oral vancomycin to reduce the incidence of Clostridioides difficile infection (CDI) in patients who suffered previous CDI and who need further hospitalization and treatment with systemic antibiotic therapy in the 90 days after the first CDI.

DETAILED DESCRIPTION:
As secondary objectives the investigators intend to:

* Evaluate the effectiveness of the treatment with oral vancomycin as part of the prophylaxis arsenal to prevent ICD in patients with previous ICD episodes stratified by the number of previous recurrences.
* Compare the severity of recurrences in both study groups.
* Compare the effectiveness of the treatment with oral vancomycin depending on the type of systemic antibiotic therapy prescribed.
* Evaluate the tolerance and the safety of the treatment with oral vancomycin in terms of secondary effects and difficulty in therapeutic compliance.
* Evaluate if the treatment with oral vancomycin has an effect in diminishing the severity of ICD recurrences.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or superior to 18 years
* Previous history of Clostridioides difficile infection in the 90 days before the study enrolment
* Need for hospitalization and need of antibiotic therapy
* Signature of informed consent

Exclusion Criteria:

* Woman of childbearing age, pregnant woman, or breastfeeding woman
* Hypersensitivity to vancomycin
* Inability to comply with study protocol
* Critically ill condition or life expectancy less than 30 days
* Patients with diagnosed inflammatory bowel disease or with any conditions that produce chronic diarrhea
* Fulfilment of the criteria for diarrhea or diagnosis of CDI at the time of assessment for eligibility or in the previous 3 days
* Therapy with oral vancomycin or any other agent with activity against C. difficile for >48 hours in the previous 3 days;.
* Prophylaxis with oral vancomycin or any other agent with activity against C. difficile within the 70 days before the assessment for eligibility
* Systemic antibiotic therapy for 72 hours or more before the recruitment
* Ongoing enrolment in another RCT evaluating the effectiveness of other drugs
* Estimated use of systemic antibiotic therapy for more than 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness of treatment with oral vancomycin in the prevention of Clostridioides difficile | 60 days after the beginning of the intervention
  Absolute difference in the rate of C. difficile infection recurrences with vancomycin Vs placebo.

SECONDARY OUTCOMES:
Effectiveness of treatment with oral vancomycin according to the number of previous recurrences | 60 days after the beginning of the intervention
  The absolute difference in the rate of C. difficile infection recurrences with vancomycin vs placebo stratified by index CDI episode (first episode or recurrence)
Effectiveness of treatment with oral vancomycin in diminishing the severity of the recurrence | 60 days after the beginning of the intervention
  The absolute difference in the rate of severe C. difficile infection recurrences with vancomycin vs placebo
Effectiveness of treatment with oral vancomycin depending on antibiotic therapy | 60 days after the beginning of the intervention
  The absolute difference in the rate of C. difficile infection recurrences with vancomycin vs placebo stratified by the type of systemic antibiotic therapy prescribed.
Tolerance and safety of treatment with oral vancomycin | 60 days after the beginning of the intervention
  Rate of major adverse events and drug-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: RAFAEL SAN-JUAN, Study Chair — HOSPITAL 12 DE OCTUBRE
Locations (1):
- Rafael San Juan, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data generated by the research will be made available as soon as possible, wherever legally and ethically possible. It is Planned to share data starting 9 months after publication, and data will be available for 24 months thereafter.
Access Criteria: IPD will be shared with investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. Proposals should be directed to rafael.san@salud.madrid.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Magill SS, Edwards JR, Bamberg W, Beldavs ZG, Dumyati G, Kainer MA, Lynfield R, Maloney M, McAllister-Hollod L, Nadle J, Ray SM, Thompson DL, Wilson LE, Fridkin SK; Emerging Infections Program Healthcare-Associated Infections and Antimicrobial Use Prevalence Survey Team. Multistate point-prevalence survey of health care-associated infections. N Engl J Med. 2014 Mar 27;370(13):1198-208. doi: 10.1056/NEJMoa1306801. PMID 24670166
- [Background] Rauseo AM, Olsen MA, Reske KA, Dubberke ER. Strategies to prevent adverse outcomes following Clostridioides difficile infection in the elderly. Expert Rev Anti Infect Ther. 2020 Mar;18(3):203-217. doi: 10.1080/14787210.2020.1717950. Epub 2020 Jan 27. PMID 31976779
- [Background] Asensio A, Monge D. [Epidemiology of Clostridium difficile infection in Spain]. Enferm Infecc Microbiol Clin. 2012 Jun;30(6):333-7. doi: 10.1016/j.eimc.2011.09.010. Epub 2011 Dec 2. Spanish. PMID 22136747
- [Background] Asensio A, Vaque-Rafart J, Calbo-Torrecillas F, Gestal-Otero JJ, Lopez-Fernandez F, Trilla-Garcia A, Canton R; EPINE Working Group. Increasing rates in Clostridium difficile infection (CDI) among hospitalised patients, Spain 1999-2007. Euro Surveill. 2008 Jul 31;13(31):18943. PMID 18761902
- [Background] McDonald LC, Owings M, Jernigan DB. Clostridium difficile infection in patients discharged from US short-stay hospitals, 1996-2003. Emerg Infect Dis. 2006 Mar;12(3):409-15. doi: 10.3201/eid1205.051064. PMID 16704777
- [Background] Eyre DW, Walker AS, Wyllie D, Dingle KE, Griffiths D, Finney J, O'Connor L, Vaughan A, Crook DW, Wilcox MH, Peto TE; Infections in Oxfordshire Research Database. Predictors of first recurrence of Clostridium difficile infection: implications for initial management. Clin Infect Dis. 2012 Aug;55 Suppl 2(Suppl 2):S77-87. doi: 10.1093/cid/cis356. PMID 22752869
- [Background] Rodriguez-Pardo D, Almirante B, Bartolome RM, Pomar V, Mirelis B, Navarro F, Soriano A, Sorli L, Martinez-Montauti J, Molins MT, Lung M, Vila J, Pahissa A; Barcelona Clostridium difficile Study Group. Epidemiology of Clostridium difficile infection and risk factors for unfavorable clinical outcomes: results of a hospital-based study in Barcelona, Spain. J Clin Microbiol. 2013 May;51(5):1465-73. doi: 10.1128/JCM.03352-12. Epub 2013 Feb 27. PMID 23447638
- [Background] Kelly CP. Can we identify patients at high risk of recurrent Clostridium difficile infection? Clin Microbiol Infect. 2012 Dec;18 Suppl 6:21-7. doi: 10.1111/1469-0691.12046. PMID 23121551
- [Background] Leav BA, Blair B, Leney M, Knauber M, Reilly C, Lowy I, Gerding DN, Kelly CP, Katchar K, Baxter R, Ambrosino D, Molrine D. Serum anti-toxin B antibody correlates with protection from recurrent Clostridium difficile infection (CDI). Vaccine. 2010 Jan 22;28(4):965-9. doi: 10.1016/j.vaccine.2009.10.144. Epub 2009 Nov 24. PMID 19941990
- [Background] Pepin J, Alary ME, Valiquette L, Raiche E, Ruel J, Fulop K, Godin D, Bourassa C. Increasing risk of relapse after treatment of Clostridium difficile colitis in Quebec, Canada. Clin Infect Dis. 2005 Jun 1;40(11):1591-7. doi: 10.1086/430315. Epub 2005 Apr 25. PMID 15889355
- [Background] Hu MY, Katchar K, Kyne L, Maroo S, Tummala S, Dreisbach V, Xu H, Leffler DA, Kelly CP. Prospective derivation and validation of a clinical prediction rule for recurrent Clostridium difficile infection. Gastroenterology. 2009 Apr;136(4):1206-14. doi: 10.1053/j.gastro.2008.12.038. Epub 2008 Dec 13. PMID 19162027
- [Background] Deshpande A, Pasupuleti V, Thota P, Pant C, Rolston DD, Hernandez AV, Donskey CJ, Fraser TG. Risk factors for recurrent Clostridium difficile infection: a systematic review and meta-analysis. Infect Control Hosp Epidemiol. 2015 Apr;36(4):452-60. doi: 10.1017/ice.2014.88. Epub 2015 Jan 28. PMID 25626326
- [Background] Cadena J, Thompson GR 3rd, Patterson JE, Nakashima B, Owens A, Echevarria K, Mortensen EM. Clinical predictors and risk factors for relapsing Clostridium difficile infection. Am J Med Sci. 2010 Apr;339(4):350-5. doi: 10.1097/MAJ.0b013e3181d3cdaa. PMID 20224312
- [Background] Ghantoji SS, Sail K, Lairson DR, DuPont HL, Garey KW. Economic healthcare costs of Clostridium difficile infection: a systematic review. J Hosp Infect. 2010 Apr;74(4):309-18. doi: 10.1016/j.jhin.2009.10.016. Epub 2010 Feb 12. PMID 20153547
- [Background] Larrainzar-Coghen T, Rodriguez-Pardo D, Puig-Asensio M, Rodriguez V, Ferrer C, Bartolome R, Pigrau C, Fernandez-Hidalgo N, Pumarola T, Almirante B. First recurrence of Clostridium difficile infection: clinical relevance, risk factors, and prognosis. Eur J Clin Microbiol Infect Dis. 2016 Mar;35(3):371-8. doi: 10.1007/s10096-015-2549-9. Epub 2016 Jan 11. PMID 26753991
- [Background] Carpenter BP, Hennessey EK, Bryant AM, Khoury JA, Crannage AJ. Identification of Factors Impacting Recurrent Clostridium difficile Infection and Development of a Risk Evaluation Tool. J Pharm Pharm Sci. 2016 Jul-Sep;19(3):349-356. doi: 10.18433/J32S41. PMID 27806252
- [Background] Zilberberg MD, Reske K, Olsen M, Yan Y, Dubberke ER. Risk factors for recurrent Clostridium difficile infection (CDI) hospitalization among hospitalized patients with an initial CDI episode: a retrospective cohort study. BMC Infect Dis. 2014 Jun 4;14:306. doi: 10.1186/1471-2334-14-306. PMID 24898123
- [Background] Aldape MJ, Rice SN, Field KP, Bryant AE, Stevens DL. Sub-lethal doses of surotomycin and vancomycin have similar effects on Clostridium difficile virulence factor production in vitro. J Med Microbiol. 2018 Dec;67(12):1689-1697. doi: 10.1099/jmm.0.000852. Epub 2018 Oct 11. PMID 30307842
- [Background] Van Hise NW, Bryant AM, Hennessey EK, Crannage AJ, Khoury JA, Manian FA. Efficacy of Oral Vancomycin in Preventing Recurrent Clostridium difficile Infection in Patients Treated With Systemic Antimicrobial Agents. Clin Infect Dis. 2016 Sep 1;63(5):651-3. doi: 10.1093/cid/ciw401. Epub 2016 Jun 17. PMID 27318333
- [Background] Cheng MP, Parkes LO, Lee TC. Efficacy of Oral Vancomycin in Preventing Recurrent Clostridium difficile Infection in Patients Treated With Systemic Antimicrobial Agents. Clin Infect Dis. 2016 Nov 15;63(10):1391-1392. doi: 10.1093/cid/ciw595. Epub 2016 Aug 27. No abstract available. PMID 27567123
- [Background] Carignan A, Poulin S, Martin P, Labbe AC, Valiquette L, Al-Bachari H, Montpetit LP, Pepin J. Efficacy of Secondary Prophylaxis With Vancomycin for Preventing Recurrent Clostridium difficile Infections. Am J Gastroenterol. 2016 Dec;111(12):1834-1840. doi: 10.1038/ajg.2016.417. Epub 2016 Sep 13. PMID 27619835
- [Background] Johnson SW, Brown SV, Priest DH. Effectiveness of Oral Vancomycin for Prevention of Healthcare Facility-Onset Clostridioides difficile Infection in Targeted Patients During Systemic Antibiotic Exposure. Clin Infect Dis. 2020 Aug 22;71(5):1133-1139. doi: 10.1093/cid/ciz966. PMID 31560051
- [Background] Bauer MP, Kuijper EJ, van Dissel JT; European Society of Clinical Microbiology and Infectious Diseases. European Society of Clinical Microbiology and Infectious Diseases (ESCMID): treatment guidance document for Clostridium difficile infection (CDI). Clin Microbiol Infect. 2009 Dec;15(12):1067-79. doi: 10.1111/j.1469-0691.2009.03099.x. PMID 19929973
- [Background] McDonald LC, Gerding DN, Johnson S, Bakken JS, Carroll KC, Coffin SE, Dubberke ER, Garey KW, Gould CV, Kelly C, Loo V, Shaklee Sammons J, Sandora TJ, Wilcox MH. Clinical Practice Guidelines for Clostridium difficile Infection in Adults and Children: 2017 Update by the Infectious Diseases Society of America (IDSA) and Society for Healthcare Epidemiology of America (SHEA). Clin Infect Dis. 2018 Mar 19;66(7):e1-e48. doi: 10.1093/cid/cix1085. PMID 29462280
- [Background] Ooijevaar RE, van Beurden YH, Terveer EM, Goorhuis A, Bauer MP, Keller JJ, Mulder CJJ, Kuijper EJ. Update of treatment algorithms for Clostridium difficile infection. Clin Microbiol Infect. 2018 May;24(5):452-462. doi: 10.1016/j.cmi.2017.12.022. Epub 2018 Jan 6. PMID 29309934
- [Background] Cornely OA, Crook DW, Esposito R, Poirier A, Somero MS, Weiss K, Sears P, Gorbach S; OPT-80-004 Clinical Study Group. Fidaxomicin versus vancomycin for infection with Clostridium difficile in Europe, Canada, and the USA: a double-blind, non-inferiority, randomised controlled trial. Lancet Infect Dis. 2012 Apr;12(4):281-9. doi: 10.1016/S1473-3099(11)70374-7. Epub 2012 Feb 8. PMID 22321770
- [Background] Johnson S, Louie TJ, Gerding DN, Cornely OA, Chasan-Taber S, Fitts D, Gelone SP, Broom C, Davidson DM; Polymer Alternative for CDI Treatment (PACT) investigators. Vancomycin, metronidazole, or tolevamer for Clostridium difficile infection: results from two multinational, randomized, controlled trials. Clin Infect Dis. 2014 Aug 1;59(3):345-54. doi: 10.1093/cid/ciu313. Epub 2014 May 5. PMID 24799326
- [Background] Louie TJ, Miller MA, Mullane KM, Weiss K, Lentnek A, Golan Y, Gorbach S, Sears P, Shue YK; OPT-80-003 Clinical Study Group. Fidaxomicin versus vancomycin for Clostridium difficile infection. N Engl J Med. 2011 Feb 3;364(5):422-31. doi: 10.1056/NEJMoa0910812. PMID 21288078
- [Background] Weiss K, Allgren RL, Sellers S. Safety analysis of fidaxomicin in comparison with oral vancomycin for Clostridium difficile infections. Clin Infect Dis. 2012 Aug;55 Suppl 2(Suppl 2):S110-5. doi: 10.1093/cid/cis390. PMID 22752858
- [Background] Charlson ME, Sax FL, MacKenzie CR, Braham RL, Fields SD, Douglas RG Jr. Morbidity during hospitalization: can we predict it? J Chronic Dis. 1987;40(7):705-12. doi: 10.1016/0021-9681(87)90107-x. PMID 3110198
- [Derived] San-Juan R, Origuen J, Campion K, Fernandez-Ruiz M, Diaz-Pollan B, Callejas-Diaz A, Candela G, Orellana MA, Lora D, Llorente Munoz I, Garcia MT, Martinez-Una M, Ferrari JM, Aguado JM. Evaluation of the effectiveness and safety of oral vancomycin versus placebo in the prevention of recurrence of Clostridioides difficile infection in patients under systemic antibiotic therapy: a phase III, randomised, double-blind clinical trial. BMJ Open. 2023 Sep 13;13(9):e072121. doi: 10.1136/bmjopen-2023-072121. PMID 37709311